CLINICAL TRIAL: NCT05927714
Title: Palatal Donor Site Wound Healing Following Periodontal Plastic Surgery Using Amnion-Chorion Membrane: Site- and Patient-Centered Outcomes
Brief Title: Palatal Donor Site Wound Healing Following Periodontal Plastic Surgery Using Amnion-Chorion Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC20230345H
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Palate; Wound
Keywords: Hemostatic agent; Amnion-chorion membrane; Accelerated wound healing; Periodontal plastic surgery
MeSH Terms: conditions — Wounds and Injuries | interventions — Hemostasis

STUDY DESIGN:
Intervention Model Description: This is a two-independent arm, parallel-design randomized, prospective trial designed to compare two standard of care techniques.
Who Masked: Participant
Masking Description: Participants will be randomly assigned to either the hemostatic agent or the amnio-chrionic membrane, but will be blinded to which standard of care intervention to which they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use Amnio Chorion Membrane (ACM) with hemostatic agent (Active Comparator): ACM or amnion-only membranes have been used in oral surgical procedures primarily because they contain a host of growth factors that play a role in normal wound healing.
  Interventions: Other: Amnion-chorion Membrane; Other: ActCel Cellulose Gauze
- Use of ActCel Cellulose Gauze (Commercial Hemostatic Agent) (Placebo Comparator): Palatal wound dressing with hemostatic agent
  Interventions: Other: ActCel Cellulose Gauze

INTERVENTIONS:
Other: Amnion-chorion Membrane — Amnio-chorion membranes specifically for palatal wound healing following free soft tissue autografts (FTSA) procedures.
  Other Names: ACM
  Arms: Use Amnio Chorion Membrane (ACM) with hemostatic agent
Other: ActCel Cellulose Gauze — When these products come in contact with blood, they convert to a gel that expands to cause direct pressure on blood vessels and control bleeding. ActCel is water-soluble and dissolves over a short time period. It can be removed easily when water, saline or hydrogen peroxide is applied.
  Other Names: Hemostatic agent

SUMMARY:
The purpose of this clinical trial is to assess if donor site healing in the palatal area and patient pain perception are similar or different when using amnio-chorion membrane (ACM) on the donor site after surgery compared to a commonly used commercial hemostatic agent (ActCel Cellulose Gauze).

DETAILED DESCRIPTION:
Resorbable oxidized cellulose materials are commonly used as hemostatic agents in medicine and dentistry. Surgicel and ActCel are used daily in surgical practice. When these products come in contact with blood, they convert to a gel that expands to cause direct pressure on blood vessels and control bleeding. ActCel is water-soluble and dissolves over a short time period. It can be removed easily when water, saline or hydrogen peroxide is applied.The study team will examine the effects of ACM as a wound dressing for the donor area and compare the rate of epithelialization with and without its use.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age 18 and 89
* Patients needing an FSTA in the area of the mouth from 2nd molar to 2nd molar in the maxilla or mandible at sites that have teeth or implants, or in sites that are edentulous
* Patients must be nonsmokers, former smokers, or current smokers who smoke <10 cigarettes per day, by self-report
* Female patients who have undergone a hysterectomy, tubal ligation, or menopause, and non- pregnant women of child-bearing potential.
* Must have access to Smartphone

Exclusion Criteria:

* Patients who disclose that they will not be able to cooperate with the follow-up schedule.
* Patients who are mentally incompetent, prisoners, or pregnant (as obtained via chart review or self-report)
* Pregnant women or women intending to become pregnant during study period
* Smokers who smoke > 10 cigarettes per day

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Wound healing time | 1, 2, 3 and 4 weeks post-operatively
  Change in Area of wound epithelialization will be measured in mm2 at 1, 2, 3 and 4 weeks postoperatively using an Early wound healing index (EHI) index. The index assesses 5 dichotomous variables, each with a "yes" or "no" assessment. "Yes" = score of 1; "No" = score of 2. Total score can range from 5 minimum to 10 maximum.
  The 5 variables are:
  * bleeding on palpation?
  * incomplete epithelialization?
  * presence of redness?
  * presence of swelling?
  * granulation tissue present?
Post-operative pain | 24, 48 and 72 hours post-surgery
  Change in pain will be assessed post surgery using a smart-phone application that captures the pain level in a scale of 1-10, where a lower number indicates a less pain

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mealey, DDS, MS, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio (Dental School), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication. IPD will all be deidentified before sharing.
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published or otherwise made available when the study is complete.